CLINICAL TRIAL: NCT01941563
Title: A Study of SI-6603 in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6603/1131; 6603/1131
Record Dates: First submitted 2013-09-04; First posted 2013-09-13 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Intervertebral Disc Disease; Lumbar Disc Disease
MeSH Terms: conditions — Intervertebral disc disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SI-6603 (Experimental): SI-6603 is administrated into the nucleus pulposus of the intervertebral disc
  Interventions: Drug: Condoliase
- Control (Sham Comparator): Sham injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Condoliase — 1.25U, intradiscal injection, one time
  Arms: SI-6603
Drug: placebo
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SI-6603 (condoliase) in patients with lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar disc herniation (L4-L5 or L5-S1) as assessed by MRI and clinical symptoms corresponding to position of the impaired nerve root.
* Patients assessed as positive in the SLR test.
* Patients with sciatica in either leg.
* Patients with no improvement from conservative treatment

Exclusion Criteria:

* Patients who have 2 or more lumbar disc herniations as assessed by MRI.
* Patients in whom a rupture into the posterior longitudinal ligament is identified by MRI.
* Patients who have received spinal injection, epidural injection, nerve block within 3 weeks prior to the time of informed consent.
* Patients who have undergone lumbar operation, or lumbar percutaneous nucleotomy or lumbar intradiscal therapies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2013-09; Primary Completion 2015-11 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Leg pain | 13 weeks
  Assessed by Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Responder rate evaluation | 13 weeks
  Assessed by leg pain (VAS), Oswestry Disability Index disability questionnaire, neurologic status (motor, sensory, reflexes), and no treatment failure

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Phoenix, Arizona
  - Gold River, California
  - Laguna Hills, California
  - Los Gatos, California
  - Murrieta, California
  - Riverside, California
  - Denver, Colorado
  - Hialeah, Florida
  - Jacksonville, Florida
  - Merritt Island, Florida
  - Miami, Florida
  - Naples, Florida
  - North Miami Beach, Florida
  - Orlando, Florida
  - Pinellas Park, Florida
  - Sarasota, Florida
  - St. Petersburg, Florida
  - Sunrise, Florida
  - Winter Park, Florida
  - Marietta, Georgia
  - Newnan, Georgia
  - Bloomington, Illinois
  - Carmel, Indiana
  - Shreveport, Louisiana
  - City of Saint Peters, Missouri
  - Hartsdale, New York
  - Eugene, Oregon
  - State College, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Sandy City, Utah
  - Edmonds, Washington